CLINICAL TRIAL: NCT03663283
Title: Liposomal Bupivacaine Interscalene Nerve Block in Shoulder Arthroplasty: A Single Blinded Prospective Randomized Control Trial
Brief Title: Liposomal Bupivacaine Interscalene Nerve Block in Shoulder Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Steven J. Hattrup, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-005366
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Arthropathy Shoulder
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacist will prepare, and dispense the medication sequentially. Medication syringes will be blinded utilizing black tape. Patients, care team in recovery, study team members collecting and recording data, and statisticians will be blinded to randomization assignment. All patients will be documented in EMR as receiving liposomal bupivacaine to ensure the blind is maintained and to ensure that safety features in the EMR for all patients receiving liposomal bupivacaine are activated. Further, all additional standard precautionary measures (e.g. wrist band) will be similarly implemented for both patient groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liposomal Bupivacaine (Experimental): Administered utilizing ultrasound guidance by an anesthesiologist. Study patients will receive 10ml (133 mg) of liposomal bupivacaine mixed with 7.5ml of 0.5% plain bupivacaine and 7.5ml of 0.25% bupivacaine. Further, 8 mg (2 ml) IV dexamethasone will be administered concomitantly at the time of the block.
  Interventions: Drug: Liposomal Bupivacaine
- Plain Bupivacaine (Active Comparator): Peripheral nerve blocks will be performed with ultrasound guidance by an anesthesiologist. Standard bupivacaine hydrochloride will be utilized. 25 ml of 0.5% bupivacaine for peripheral nerve block will be utilized. Further, 8 mg (2 ml) IV dexamethasone will be administered concomitantly at the time of the block.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Liposomal Bupivacaine — Interscalene Nerve Blocks
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine Hydrochloride — Interscalene Nerve Blocks
  Arms: Plain Bupivacaine

SUMMARY:
The objective of this study is to determine if peripheral nerve block with liposomal bupivacaine in combination with standard bupivacaine will prolong the duration of block, improve pain scores, and decrease opioid utilization in the post-operative period when compared to peripheral nerve block with standard bupivacaine alone.

DETAILED DESCRIPTION:
This is a prospective, single-blinded randomized clinical trial comparing outcomes in patients undergoing total shoulder arthroplasty (anatomic and reverse) who receive a peripheral nerve block with liposomal bupivacaine in combination with standard bupivacaine versus standard bupivacaine alone. Once consent is obtained, baseline characteristics will be recorded and patients will be randomized to intervention or control. Following surgery, patients will be followed until their 3-week post-operative visit. The primary outcome measure will be the mean difference in patient pain scores over the first 72 hours post-operatively between two groups. Secondary outcomes will include: (1) Total opioid consumption (as measured utilizing morphine intravenous equivalents) in first 72 hours and at 3 weeks (2) Patient perceived duration of block determined as the time patient perceives complete resolution of block (3) Patient satisfaction with pain control at 72 hours, 3 weeks post-operatively and patient reported outcome measures (SANE, SST, ASES, VR-12) at 3 weeks post-operatively.

ELIGIBILITY:
Inclusion Criteria

* All adult patients (>18 years of age)
* Patients undergoing standard or reverse total shoulder arthroplasty for the primary diagnoses of glenohumeral arthritis or cuff tear arthropathy
* Cognitively intact with the ability to give informed consent as outlined by our institutional review board.
* Patients must be capable of participating in the post-operative electronic survey and / or able to maintain a written diary of events

Exclusion Criteria

* Non-elective cases
* Infection, tumor, trauma
* Weight < 50 kg
* Patients with any contraindications to regional anesthesia including allergy or hypersensitivity to amide-type local anesthetics
* Patients with allergy to any component of medication regimen e.g. amide- type local anesthetics, oxycodone, hydromorphone, fentanyl
* Chronic pain patients with history of chronic opioid use (defined as 20 mg morphine equivalent / day for greater than 30 days pre-operatively
* Concurrent painful physical condition that may require analgesic treatment that is not related to the shoulder surgery (chronic peripheral neuropathy, radiculopathy, or other neurologic disorder)
* Severe hepatic disease defined by clinical evidence of liver disease with abnormal liver function tests.
* Pregnancy
* Respiratory disease that contraindicates interscalene nerve block (elevated contralateral hemidiaphragm, contralateral pneumonectomy, or severe COPD with FEV1 < 50% predicted, and 02 dependence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Hattrup, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials
- See also: PubMed — https://pubmed.ncbi.nlm.nih.gov/33045330/

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine: Administered utilizing ultrasound guidance by an anesthesiologist. Study patients received 10ml (133 mg) of liposomal bupivacaine mixed with 7.5ml of 0.5% plain bupivacaine and 7.5ml of 0.25% bupivacaine. Further, 8 mg (2 ml) IV dexamethasone was administered concomitantly at the time of the block.
  Liposomal Bupivacaine: Interscalene Nerve Blocks
- Plain Bupivacaine: Peripheral nerve blocks were performed with ultrasound guidance by an anesthesiologist. Standard bupivacaine hydrochloride was utilized. 25 ml of 0.5% bupivacaine for peripheral nerve block was utilized. Further, 8 mg (2 ml) IV dexamethasone was administered concomitantly at the time of the block.
  Bupivacaine Hydrochloride: Interscalene Nerve Blocks
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine
Started | 52 | 52
Completed | 52 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (6.84) | 69.2 (10.15) | 69.6 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 30 | 28 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Patient Pain Scores
Description: Patient pain scores over the first 72 hours post-operatively as measured by the Visual Analogue Scale where Zero represents no pain and ten represents severe pain.
Time Frame: 72 hours post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine
Number analyzed (Participants) | 52 | 52
score on a scale | 4.0 (2.57) | 2.8 (1.88)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Plain Bupivacaine; Test type: Superiority; p = .0197, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Opioid Consumption
Description: Total opioid consumption as measured by morphine milligram equivalent (MME) in first 72 hours and at 3 weeks
Time Frame: Measured at 72 hours and at 3 weeks post-operatively
Measure: Mean (Standard Deviation); unit: morphine milligram equivalent (MME)
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine
Number analyzed (Participants) | 52 | 52
morphine milligram equivalent (MME)
  72 hours | 45.6 (37.55) | 56.2 (35.43)
  3 weeks | 133.9 (110.52) | 150.9 (138.4)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Plain Bupivacaine; 72 hours; Test type: Superiority; p = 0.584, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Liposomal Bupivacaine vs Plain Bupivacaine; 3 weeks; Test type: Superiority; p = .5800, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Time to Cessation of Nerve Blockade
Description: Measured by the number of subjects who reported cessation of nerve blockade as the first reported postoperative pain score of 3 or greater at the surgical site.
Time Frame: 4, 8, 12, 16, 20, 24, and 28 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine
Number analyzed (Participants) | 47 | 45
Participants
  4 hours | 16 | 12
  8 hours | 31 | 19
  12 hours | 38 | 28
  16 hours | 43 | 35
  20 hours | 43 | 41
  24 hours | 46 | 44
  28 hours | 47 | 45
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Plain Bupivacaine; Test type: Superiority; p = 0.11, Log Rank

4. Secondary Outcome: Satisfaction With Pain Control Using Satisfaction Scale
Description: Patient satisfaction with pain control at 72 hours post-operatively and three weeks post operatively using Patient Satisfaction with Pain Management Pain Scale where Zero represents unsatisfactory pain management and ten represents perfect pain management.
Time Frame: Measured at 72 hours and at three weeks post-operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine
Number analyzed (Participants) | 52 | 52
units on a scale
  72 hours | 6.6 (2.74) | 6.9 (2.64)
  3 weeks | 7.5 (2.52) | 7.8 (2.23)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Plain Bupivacaine; 72 hours; Test type: Superiority; p = .7018, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Liposomal Bupivacaine vs Plain Bupivacaine; Week 3; Test type: Superiority; p = .5327, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to treatment follow up visit, approximately 10 days.
Arm/Group | Liposomal Bupivacaine | Plain Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT03663283/Prot_SAP_000.pdf